CLINICAL TRIAL: NCT03983642
Title: Effects of the Nintendo Wii Fit Game Training on Balance Among Lebanese Elderly
Brief Title: Effects of the Nintendo Wii Fit Game Training on Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese German University (Other)
Responsible Party: Principal Investigator, Mohammed Ali FAKHRO, DPT, Coordinator, Lebanese German University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Effects of Nintendo Wii Fit
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Balance; Distorted
Keywords: Dynamic balance; Static balance; Wii Fit; Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received a session of 40min for an 8 weeks' period. Both games requested the participants to stand on a balance board in front of the television, without shoes, while trying to control their avatars by shifting their body weights.
  Interventions: Device: Wii balance board
- Control group (No Intervention): Participants in the control group were followed-up by an assessor, who made sure that they will not get involved in any type of training program during the eight weeks' period of the trial.

INTERVENTIONS:
Device: Wii balance board — Numerous video games exist to interact with the Wii Balance Board. One game that has been used in prior balance studies is Wii Fit.
  On the first 4 weeks, balance training started with "Soccer Heading" game. The participants were asked to control their avatar by leaning to left or to the right in order to avoid the objects that were thrown towards them, and try to score the balls inside the net. The participants performed 3 sets of 5 rounds (2min each), totaling 30 min, and rested for 1 min between each set.
  "Table Tilt" game continued for the remaining 4 weeks. Participants tried to enter balls into the holes by shifting their body weight on the balance board causing it to tilt in all directions. This game was divided into multiple levels of 30 seconds each, repeated over 30 min, with a one-minute rest interval between every 10 minutes of training. Moreover, 20 extra seconds were added each time a participant has won a level.
  Arms: Intervention group

SUMMARY:
This study is a single-blinded prospective longitudinal randomized controlled trial (RCT). The experiment took place over a period of eight weeks. Elderly participants were randomized into two groups (intervention and control). Participants of each group were followed-up carefully by assessors over three times per week, for a total of 24 sessions and during the data collection periods as well. Dynamic and static balance measures were compared between the groups on two occasions (baseline, and post-test). Timed Up and Go (TUG) test, and the Nintendo Wii Balance Board (NWBB) were used to measure the dynamic and static balance respectively.

DETAILED DESCRIPTION:
Design

This study embraced an experimental randomized controlled trial (RCT) design, where both baseline and post-test measures were recorded for both the dynamic and static balance. Ethical approval was obtained from the Lebanese German University Institutional Review Board. Every participant in this study received an information sheet which contains sections on (a) research purpose, (b) voluntary participation, (c) study protocol, (d) risks and benefits, (e) confidentiality, and (f) contact personals.

Participants and Selection Criteria

After a random selection of both of Tyre and Saida districts to represent the South governorate (cluster sampling), all the geriatric centers present in these areas were included in the study.

Participants inclusion criteria included (a) age of 65 years and above, (b) impaired dynamic balance characterized by TUG test score >14 seconds, (c) Montreal Cognitive Assessment (MoCA) test score ≥ 23, (d)good vision, and (e) no vestibular disorders. On the other hand, (a) those who were on a wheelchair or used walkers for mobility, (b) sustained a fracture or underwent orthopedic surgery to the lower extremities within the last 6 months, and (c) have an amputated limb, were excluded. After applying the inclusion and exclusion criteria, 64 participants remained and accepted to enroll in the study. Four of these participants dropped -out eventually, three from the intervention group, and one from the control group, leaving these two groups equally split.

Data Collection Methods

In order to collect the data of the study variables, TUG test and Nintendo Wii Balance Board (NWBB) were used to measure balance-related outcomes. Whereas, the MoCA test was used to screen for cognitive impairment.

At the moment of data collection, the assessor was blind to the group to which the participants belonged. In addition, this assessor was not involved in the implementation of the study protocol.

Timed Up and Go (TUG) test.

The TUG test is a simple yet effective test that assesses a person's balance in mobility. The participant is asked to sit on a chair, rise up, walk three meters, turn around and return to sit on the chair. The time was measured using a stopwatch in seconds. Normative values for age groups were as follows: (a) 60-69 years between 7.1 - 9.0 seconds; b) 70-79 years between 8.2 - 10.2 seconds; and c) 80-99 years between 10.0 - 12.7 seconds. Participants who finished with a score above 14 seconds were associated with high risks of falls.

Intratester and intertester reliability have been reported as high in elderly populations (ICC = 0.92-0.99).

Nintendo Wii Balance Board (NWBB).

Compared to inanimate objects, the human body has the ability to control stability and modulate body posture when the vertical projection of the center of mass (COM) approaches Base of Support (BOS). These abilities emerge from a complex interaction between the musculoskeletal and afferent/efferent neural systems, and the central nervous system processing, often collectively termed as "postural control". Postural control was defined as: "the act of maintaining, achieving or restoring a state of balance during any posture or activity". The specific demand of the postural control system in a given situation is dependent upon the task being done, the individual's abilities and the environment.

Moreover, laboratory-based assessment using measures center of pressure (COP) recorded from a force platform (FP) is considered the gold standard measure of balance. COP may serve as an objective and pragmatic outcome measure derived from the postural control system. The COP position represents the location of the resultant Center of gravity. The FP technique is sensitive, objective and quantitative, however unfortunately also expensive, highly immobile and often technically difficult to carry out and subsequently process. For these reasons, more simple and integrative measures are needed in large scale clinical patient settings.

The NWBB is an easy-to-use, portable and low-cost force platform instrumented with sensitive force sensors positioned in each corner. Good-to-excellent test-retest reproducibility has been demonstrated during static bilateral stance. Similarly, the inter-rater reliability (ICC: 0.79-0.89) was considered high in terms of COP path length and COP velocity. In addition, good-to-excellent concurrent validity was observed when COP recordings based on the NWBB were compared to similar data obtained using an FP (AMTI model).

The NWBB (Nintendo, Kyoto, Japan), is a 26 cm× 44 cm rigid platform with four uni-axial vertical force transducers located in the feet at the corners of the board, one transducer per foot. Each transducer is a load cell consisting of a metal bar with a strain gauge that converts applied force to a voltage that is digitized and transmitted wirelessly by electronics in the NWBB. Participants were instructed to stand still while adopting their usual posture on the platform for 30 seconds. To collect data from the NWBB, data was streamed to a computer (Lenovo, Windows 10) using the Bluetooth Human Interface Device (HID) wireless protocol and custom programs written in Java (Oracle) and Matlab (Mathworks, Natick, MA). Computer analysis of COP displacements recorded percentage of distribution of the COP between the left and right legs. If the percentage was not equally distributed between the two legs, this indicated an impaired balance, and that COM was outside the BOS.

Numerous video games exist to interact with the Wii Balance Board. One game that has been used in prior balance studies is Wii Fit. This game allowed users to complete various training modes such as yoga, strength training, aerobics, and balance games. These training modes are similar to traditional balance training interventions but provide real-time force feedback. Among the games that target balance and were chosen for this study were the (a) Soccer Heading, and (b) Table-tilt games.

Montreal Cognitive Assessment (MoCA) test.

The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It is a brief (30-question) test that takes around 10 to 12 minutes to administer. The MoCA evaluates different types of cognitive abilities, which include (a) short-term memory (5 points, (b) visuospatial abilities (4 points), (c) executive functioning (4 points), (d) attention, concentration, and working memory (6 points), (e) language (5 points), and (f) orientation to time and place (6 points).

The MoCA is scored by adding the total scores of items and the authors stated that a clinical cutoff score of 26 or above was to be considered normal. The MoCA was influenced by education, prompting the authors to recommend adding one point to the cut score for elders with over 12 years of education.

In the original validation study, the MoCA outperformed the Mini-Mental State Examination (MMSE) across both mild cognitive impairment (MCI) and Alzheimer disease groups (AD) (MoCA sensitivity 0.90 and 1.00, respectively), but its specificity was observed to be lower than that of the MMSE (although still high at 0.87). Positive predictive value (PPV) for the MoCA was 0.89 for both groups and negative predictive value (NPV) of 0.91 and 1.00 for the MCI and AD groups, respectively.

Subsequent studies have demonstrated a trend characterized by high sensitivity and low specificity for the MoCA. At a cutoff of 26, the MoCA yielded high sensitivity but low specificity, however, when a cut score of 23 was used, both sensitivity and specificity were excellent (0.96 and 0.95, respectively).

The MoCA is a promising alternative to the MMSE because of its sensitivity to the early detection of dementia and MCI.

Procedure

In order to recruit the participants, geriatric specialized centers were visited across the regions of Saida and Tyre districts. Eligible elderly participants signed an informed consent to participate and then were randomized by a mean of a randomization site (https://www.randomizer.org/) to two groups. The intervention group received the Wii Fit balance training, while the control group received no training. Both groups were gender matched.

The experiment was conducted over a period of eight weeks. The MoCa test was performed to enroll eligible participants in the study (score ≥ 23). Afterward, the TUG, NWBB tests were applied twice, at the beginning of the trial (baseline data), and at the end of the trial to compare the measures. Participants of the intervention group were followed-up carefully by assessors during their intervention sessions three times a week, for a total of 24 sessions and during data collection.

Intervention group.

The intervention group received a balance training session that took 40 minutes to complete (five minutes for warm up, 30 minutes for balance training, and five minutes for cooldown). Balance training started at the beginning of the first four weeks, with the "Soccer Heading" game. This game was considered easier than the "Table Tilt" game that began continued at the remaining four weeks.

The Soccer Heading game requested the participant to stand on a balance board in front of the television, without shoes, while soccer balls and other objects are thrown towards the participant. The participant was asked to control his avatar by leaning to left and to the right in order to avoid the objects and score the balls inside the net, challenging both dynamic postural control and coordination. Each round is made up of two minutes. The participants performed 3 sets of five rounds, totaling 30 minutes. The participant rested for one minute between each set.

The Table Tilt game requested the participant to stand on the balance board in front of the television, without shoes, and he/she was asked to enter the ball (s) into the hole (s) while maneuvering a floating table by shifting the body weight on the balance board causing it to tilt (in all direction). The participant should also pay attention not to drop the ball (s) out of the floating board. The game was divided into multiple levels, where each level duration was 30 seconds. After the participants had won a level, an extra 20 seconds was added. The game was repeated over a period of 30 minutes, with a one-minute rest interval every 10 minutes.

Control group.

Participants in the control group were followed-up by an assessor, who made sure that they will not get involved in any type of training program during the eight weeks' period of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. age of 65 years and above,
2. impaired dynamic balance characterized by TUG test score >14 seconds,
3. Montreal Cognitive Assessment (MoCA) test score ≥ 23,
4. good vision,
5. no vestibular disorders.

Exclusion Criteria:

1. those who were on a wheelchair or used walkers for mobility,
2. sustained a fracture or underwent orthopedic surgery to the lower extremities within the last 6 months,
3. have an amputated limb.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) test- Change | "Baseline and after 8 weeks"
  The TUG test is a simple yet effective test that assesses a person's balance in mobility. The participant is asked to sit on a chair, rise up, walk three meters, turn around and return to sit on the chair. The time was measured using a stopwatch in seconds. Normative values for age groups were as follows: (a) 60-69 years between 7.1 - 9.0 seconds; b) 70-79 years between 8.2 - 10.2 seconds; and c) 80-99 years between 10.0 - 12.7 seconds. Participants who finished with a score above 14 seconds were associated with high risks of falls (Bohannon, 2006).
  Intratester and intertester reliability have been reported as high in elderly populations (ICC = 0.92-0.99) (Steffen, Hacker, & Mollinger, 2002).
Nintendo Wii Balance Board (NWBB)- Change | "Baseline and after 8 weeks"
  The NWBB (Nintendo, Kyoto, Japan), is a 26 cm× 44 cm rigid low-cost force platform with four uni-axial vertical force transducers located in the feet at the corners of the board, one transducer per foot. Each transducer is a load cell consisting of a metal bar with a strain gauge that converts applied force to a voltage that is digitized and transmitted wirelessly by electronics in the NWBB (Ogasawara, 2012). To collect data from the NWBB, data was streamed to a computer (Lenovo, Windows 10) using the Bluetooth HID wireless protocol and custom programs written in Java (Oracle) and Matlab (Mathworks, Natick, MA).
  Good-to-excellent test-retest reproducibility has been demonstrated during static bilateral stance (Clark et al., 2010). Similarly, the inter-rater reliability (ICC: 0.79-0.89) was considered high in terms of COP path length and COP velocity (Ogasawara, 2012). In addition, good-to-excellent concurrent validity was observed (Clark et al, 2010).

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) test | "Baseline"
  The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It is a brief (30-question) test that takes around 10 to 12 minutes to administer. MoCA evaluates different types of cognitive abilities (Nasreddine et al., 2005).
  MoCA is scored by adding the total scores of items and the authors stated that a clinical cutoff score of 26 or above was to be considered normal. It was influenced by education, prompting the authors to recommend adding one point to the cut score for elders with over 12 years of education (Nasreddine et al., 2005). Subsequent studies have demonstrated a trend characterized by high sensitivity and low specificity for the MoCA. At a cutoff of 26, the MoCA yielded high sensitivity but low specificity, however, when a cut score of 23 was used, both sensitivity and specificity were excellent (0.96 and 0.95, respectively) (Luis, Keegan, & Mullan, 2009).

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese German University, Jounieh, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: No